CLINICAL TRIAL: NCT05311137
Title: Application of the Closed-loop Treatment Concept of Atrial Fibrillation in the Atrial Fibrillation Population in the Northern Shanghai Community
Brief Title: Study of the Closed-loop Treatment Concept of Atrial Fibrillation in the Atrial Fibrillation Population
Acronym: CONTROL-AF
Status: Recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Director, Director of Cardiovascular Medicine, Shanghai 10th People's Hospital
Other Study IDs: CONTROL-AF
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation；closed-loop treatment；
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation; Cryosurgery; Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Closed-loop Group: Groups of Patients Adhering to Closed-Loop Therapy.
  Interventions: Procedure: Radiofrequency ablation
- No Closed-loop Group: Patients who have not undergone closed-loop treatment or patients who have not undergone standard surgery and medication.
- Exchange Group: Groups of patients with delayed compliance with closed-loop therapy for atrial fibrillation.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Combined use of radiofrequency ablation, cryoablation, left bundle branch pacing, and left atrial appendage closure according to the actual situation of the patient.
  Other Names: cryoablation;; left bundle branch pacing;; left atrial appendage occlusion;
  Groups: Closed-loop Group; Exchange Group

SUMMARY:
This study aims to evaluate the concept of closed-loop treatment of atrial fibrillation for the optimization of the treatment strategy.

DETAILED DESCRIPTION:
This study aims to evaluate the concept of closed-loop treatment of atrial fibrillation for the optimization of the treatment strategy, the improvement of disease outcome and the economic value of the atrial fibrillation population in the northern Shanghai community. Improve the disease cognition of patients with atrial fibrillation, and promote the development of the concept of closed-loop treatment of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation patients；Ability to act autonomously, understand and sign informed consent；

Exclusion Criteria:

* none（All patients with atrial fibrillation were enrolled in this study indiscriminately and followed up）

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation patients in North Shanghai area.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | 2 years
  The recurrence of atrial fibrillation and the degree of burden of atrial fibrillation in patients.
Heart failure | 5 years
  Degree of heart failure (including EF%, NYHA score, etc.)
Stroke | 5 years
  stroke attack(Check for new cerebral infarction by MRI）

SECONDARY OUTCOMES:
bleeding | 2 years
  major bleeding event
Cardiovascular MACE events | 5 years
  Cardiovascular MACE events

CONTACTS AND LOCATIONS:
Overall Officials: WeiYa Xu, PhD, Study Chair — No. 301 Yanchang Middle Road, Jing'an District, Shanghai, China
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No